CLINICAL TRIAL: NCT05149573
Title: Investigation of Non-Invasive Pulsed Electromagnetic Field (PEMF) Therapy for Female Patients With Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS)
Brief Title: Investigation of PEMF Therapy for Female Patients With IC/BPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00079006; 1R01DK128233-01A1 (NIH)
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-08

CONDITIONS: Interstitial Cystitis; Chronic Interstitial Cystitis; Bladder Pain Syndrome
Keywords: interstitial cystitis; bladder pain syndrome; painful bladder syndrome; painful bladder; bladder pain; urinary urgency; urinary frequency; pulsed electromagnetic field
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Intervention Model Description: This study is designed as a double-blind, sham-controlled clinical trial separated into two Aims. Aim 1 will include 60 female adults with IC/BPS, divided into two groups: 1) 30 participants with an anesthetic bladder capacity (BC) ≤ 400cc and 2) 30 participants with BC > 400cc. Patients within each of the two groups will be randomly assigned in a 1:1 ratio to either the PEMF (treatment) or Sham (control) group. The Sham device is identical to the treatment device but does not deliver PEMF. All participants will be instructed to use their device every day, morning and evening, for 8-minute sessions over a 4-week period.
  Aim 2 will include an additional cohort of 15 female adults with IC/BPS. These participants will undergo the standard 4-week regimen of PEMF therapy, followed by a one-week-per-month maintenance period of twice daily PEMF therapy for an additional 3 months post-enrollment (the fourth week in months 2, 3, and 4).
Who Masked: Participant, Investigator
Masking Description: The participant and study investigator will not know whether the study participant has received PEMF (treatment) or Sham (control) therapy. Only the study coordinator, who will distribute the devices to study participants, will be unmasked to the therapies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- 4-Week Treatment with no Maintenance Period (Active Comparator): Treatment will be provided via self-administration of pulsed electromagnetic field (PEMF) therapy using the B. Body (full body mat) and B. Pad (targeted pelvic pad). The participant will lie the B. Body mat on any flat surface and lay on the mat with the smaller B. Pad placed directly over the pelvic area. The PEMF device (attached to the control unit) has been pre-programmed to deliver the same level of energy every time. Participants will be instructed to administer this home treatment twice a day (morning and evening) for 8-minute sessions over a 4-week period. After 4 weeks, participants will return the device and complete one set of electronic questionnaires during the last week of the month for the following 3 months.
  Interventions: Device: Pulsed Electromagnetic Field (PEMF) Device
- 4-Week Sham Treatment with no Maintenance Period (Sham Comparator): Participants will be provided with a sham B. Body and B. Pad that appears identical to the active pulsed electromagnetic field (PEMF) device. The participant will lie the sham B. Body mat on any flat surface and lay on the mat with the smaller sham B. Pad placed directly over the pelvic area. The participant will be instructed to administer this sham treatment twice a day (morning and evening) for 8-minute sessions over a 4-week period. After 4 weeks, participants will return the sham device and complete one set of electronic questionnaires during the last week of the month for the following 3 months.
  Interventions: Device: Sham Pulsed Electromagnetic Field (PEMF) Device
- 4-Week Treatment with 1-Week-Per-Month Maintenance Period for an Additional 3 Months (Active Comparator): Treatment will be provided via self-administration of pulsed electromagnetic field (PEMF) therapy using the B. Body (full body mat) and B. Pad (targeted pelvic pad). The participant will lie the B. Body mat on any flat surface and lay on the mat with the smaller B. Pad placed directly over the pelvic area. The PEMF device (attached to the control unit) has been pre-programmed to deliver the same level of energy every time. Participants will be instructed to administer this home treatment twice a day (morning and evening) for 8-minute sessions over a 4-week period. After 4 weeks, participants will keep the device and use it for 1 week (7 days) during the last week of the month for the following 3 months. Each participant in this group will be asked to complete a set of electronic questionnaires immediately following their week-long maintenance treatment during the last 3 months of the study.
  Interventions: Device: Pulsed Electromagnetic Field (PEMF) Device

INTERVENTIONS:
Device: Pulsed Electromagnetic Field (PEMF) Device — BEMER PEMF device consists of a B. Body (full body mat), B. Pad (targeted pelvic pad), and Control Unit which powers the device. Both B. Body and B. Pad must be plugged in simultaneously into the Control Unit and activated individually. B. Body must be placed on a flat surface (e.g. floor, bed, reclining chair, etc) for best results.
  Other Names: BEMER PEMF; BEMER B. Body; BEMER B. Pad; BEMER Control Unit
  Arms: 4-Week Treatment with 1-Week-Per-Month Maintenance Period for an Additional 3 Months; 4-Week Treatment with no Maintenance Period
Device: Sham Pulsed Electromagnetic Field (PEMF) Device — The sham PEMF device appears identical to the BEMER PEMF device, with all of the same components and accessories, but does not emit a pulsed electromagnetic field.
  Arms: 4-Week Sham Treatment with no Maintenance Period

SUMMARY:
The purpose of this study is to gather information about the safety and effectiveness of the non-pharmacological (non-drug), non-invasive treatment known as low-frequency pulsed electromagnetic field (PEMF) therapy. The study team will distribute the PEMF device to female adults with Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS) to measure its ability to decrease bladder and pelvic pain as well as other urinary symptoms associated with IC/BPS. There are two sequential Aims in this study and subjects will be recruited to participate in only one Aim. In both Aims, data will be collected at baseline/enrollment, 4-weeks after using PEMF therapy, and 8, 12, and 16 weeks post-enrollment.

DETAILED DESCRIPTION:
Interstitial cystitis/bladder pain syndrome (IC/BPS) is a clinical diagnosis based primarily on chronic symptoms of pain perceived by the patient to emanate from the bladder and/or pelvis associated with urinary urgency or frequency in the absence of another identifiable cause of the symptoms. Although it is not a life-threatening disease, the chronicity and severity of pain, along with other urinary symptoms, causes great impairment in a patient's quality of life. In addition, IC/BPS poses a significant clinical challenge for many reasons. For one, the pathophysiology described in the literature is incompletely determined and likely multi-factorial, including factors such as inflammation, neurovascular dysfunction, ion imbalance, and impaired urothelial cell integrity. Consequently, there are many options for IC/BPS therapy, many of which are driven primarily by patient-reported symptoms. In this regard, IC/BPS patients with moderate to severe pain typically require multi-modal therapy, often resulting in incomplete or no resolution of symptoms. Another clinical challenge is the heterogeneity of the symptoms. While pelvic pain is the distinguishing characteristic, patients with IC/BPS also routinely present with additional urological and non-urological medical symptoms and syndromes. This has led to the description of two specific sub-phenotypes in IC/BPS based on anesthetized bladder capacity (BC), in which patients with BC < 400 cc are more likely to experience severe pain, urgency and frequency (bladder centric sub-phenotype), and patients with BC > 400 cc (non-bladder centric sub-phenotype) have a higher prevalence of non-urological associated syndromes (NUAS) such as fibromyalgia, chronic fatigue symptoms, irritable bowel syndrome, endometriosis and sicca syndrome.

Pulsed Electromagnetic Field (PEMF) therapy may present a promising alternative therapy for patients with IC/BPS. PEMF is a safe, non-invasive, and effective therapy currently used for wound healing, bone-related diseases (osteoarthritis, rheumatoid arthritis), and chronic pain states (chronic lower back pain, fibromyalgia), the latter of which are frequently associated with IC/BPS as NUAS. Based on Faraday's law, electromagnetic interactions (e.g. PEMF) with biological processes and conditions (e.g. IC/BPS) will theoretically address many of the proposed pathophysiological causes of the condition. While the mechanism(s) of action are not fully understood, PEMF therapy has been shown in several studies (randomized, double-blinded, placebo-controlled trials) to decrease the output of pro-inflammatory proteins, improve oxygenation of blood and tissue, stabilize transmembrane action potential and ion channels, and stimulate tissue regeneration. Thus, PEMF may provide a safe, non-invasive therapeutic option that would be complementary to, or serve as an alternative for, the treatments that are currently being administered in IC/BPS for pain reduction. Of note, PEMF has demonstrated an excellent safety profile with no associated systemic risks reported to date. Additionally, the application of exogenous PEMF to stimulate the pelvic floor muscle has recently been introduced for treating urge and/or stress urinary incontinence and overactive bladder. Furthermore, if patient safety and efficacy for pain reduction are demonstrated, these feasibility studies will provide the foundation for larger multi-site trials to determine additional parameters regarding the appropriate number of treatments as well as the duration of benefit (pain relief) following treatments.

The purpose of this study is to determine the safety and efficacy of PEMF therapy to significantly reduce pain among female patients with IC/BPS (Aim 1) and to evaluate the duration of benefit from PEMF therapy with and without maintenance treatments over a 4-month period (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* Previously established clinical diagnosis of IC/PS
* Current numeric rating scale (NRS) score of ≥ 6
* History of cystoscopy with hydrodistension with bladder capacity determination under anesthesia
* No cognitive deficits

Exclusion Criteria:

* History of bladder, ovarian, vaginal cancer
* History of urethral diverticulum
* History of radiation cystitis
* History of spinal cord injury or spina bifida
* History of Parkinson's disease, multiple sclerosis, or stroke
* Current placement of a pacemaker or metal prosthesis
* Active urinary tract infection
* BMI > 40
* Residual urine of > 100cc
* Current pregnant

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Subject must be biologically Female
Enrollment: 75 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Pelvic pain, as measured by the Brief Pain Inventory (BPI) Short Form | Baseline
  The BPI Short Form is a validated questionnaire to assess the severity of systemic and pelvic pain and its interference in overall quality of life. Pain severity is measured through four 11-point numeric rating scales (NRS) assessing pain at its "worst," "least," and "average," within the past week, and pain "right now" (at the time of short form completion), with the composite (mean score) of all four scales indicating overall pelvic pain. Pain interference is measured through 7 scales, with scores ranging from 0 (does not interfere) to 10 (completely interferes), for different daily activities. The composite score for the interference items is used to assess overall pain interference, with higher scores indicating greater symptom severity and a change in 2 points indicating a significant change in pain. The form also consists of 3 pain body maps to identify specific locations of pain, and 2 questions related to the effect of current medications on pain.
Change from baseline pelvic pain, as measured by the Brief Pain Inventory (BPI) Short Form | Week 4
  The BPI Short Form is a validated questionnaire to assess the severity of systemic and pelvic pain and its interference in overall quality of life. Pain severity is measured through four 11-point numeric rating scales (NRS) assessing pain at its "worst," "least," and "average," within the past week, and pain "right now" (at the time of short form completion), with the composite (mean score) of all four scales indicating overall pelvic pain. Pain interference is measured through 7 scales, with scores ranging from 0 (does not interfere) to 10 (completely interferes), for different daily activities. The composite score for the interference items is used to assess overall pain interference, with higher scores indicating greater symptom severity and a change in 2 points indicating a significant change in pain. The form also consists of 3 pain body maps to identify specific locations of pain, and 2 questions related to the effect of current medications on pain.
Change from baseline pelvic pain, as measured by the Brief Pain Inventory (BPI) Short Form | Week 8
  The BPI Short Form is a validated questionnaire to assess the severity of systemic and pelvic pain and its interference in overall quality of life. Pain severity is measured through four 11-point numeric rating scales (NRS) assessing pain at its "worst," "least," and "average," within the past week, and pain "right now" (at the time of short form completion), with the composite (mean score) of all four scales indicating overall pelvic pain. Pain interference is measured through 7 scales, with scores ranging from 0 (does not interfere) to 10 (completely interferes), for different daily activities. The composite score for the interference items is used to assess overall pain interference, with higher scores indicating greater symptom severity and a change in 2 points indicating a significant change in pain. The form also consists of 3 pain body maps to identify specific locations of pain, and 2 questions related to the effect of current medications on pain.
Change from baseline pelvic pain, as measured by the Brief Pain Inventory (BPI) Short Form | Week 12
  The BPI Short Form is a validated questionnaire to assess the severity of systemic and pelvic pain and its interference in overall quality of life. Pain severity is measured through four 11-point numeric rating scales (NRS) assessing pain at its "worst," "least," and "average," within the past week, and pain "right now" (at the time of short form completion), with the composite (mean score) of all four scales indicating overall pelvic pain. Pain interference is measured through 7 scales, with scores ranging from 0 (does not interfere) to 10 (completely interferes), for different daily activities. The composite score for the interference items is used to assess overall pain interference, with higher scores indicating greater symptom severity and a change in 2 points indicating a significant change in pain. The form also consists of 3 pain body maps to identify specific locations of pain, and 2 questions related to the effect of current medications on pain.
Change from baseline pelvic pain, as measured by the Brief Pain Inventory (BPI) Short Form | Week 16
  The BPI Short Form is a validated questionnaire to assess the severity of systemic and pelvic pain and its interference in overall quality of life. Pain severity is measured through four 11-point numeric rating scales (NRS) assessing pain at its "worst," "least," and "average," within the past week, and pain "right now" (at the time of short form completion), with the composite (mean score) of all four scales indicating overall pelvic pain. Pain interference is measured through 7 scales, with scores ranging from 0 (does not interfere) to 10 (completely interferes), for different daily activities. The composite score for the interference items is used to assess overall pain interference, with higher scores indicating greater symptom severity and a change in 2 points indicating a significant change in pain. The form also consists of 3 pain body maps to identify specific locations of pain, and 2 questions related to the effect of current medications on pain.

SECONDARY OUTCOMES:
Change in Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS) symptoms, as measured by O'Leary Sant Interstitial Cystitis Symptom Index and Problem Index (ICSI/ICPI) | Baseline, Week 4, Week 8, Week 12, and Week 16
  The ICSI (score range: 0-19 points) and ICPI (score range: 0-16 points) contain four questions related to urinary and pain symptoms. For the symptoms index, 3 of the 4 questions utilize a range of 0-5 with 0 indicated the symptom is never experienced and 5 indicating the symptom is almost always experienced. The fourth question utilizes a range of 0-4 with 0 indicating the symptom is never experienced and 4 indicating the symptom is almost always experienced. For the problem index, all four questions utilize a range of 0-4 with 0 indicating it is no problem and 4 indicating it is a big problem.
Change in Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS) symptoms, as measured by Pelvic Pain and Urgency/Frequency (PUF) Patient Symptom Scale | Baseline, Week 4, Week 8, Week 12, and Week 16
  The PUF Patient Symptom Scale is a validated instrument used to assess the severity of symptoms associated with IC/BPS and the degree to which these symptoms "bother" a patient. It is separated into two subsections, scored individually as the Symptom Score and Bother Score, to produce one composite score. The symptom score is comprised of 7 items addressing urinary frequency, urgency, nocturia, dyspareunia, and pelvic pain. Each question is scored from 0 (never) to 3 (always) or 1 (mild) to 3 (severe), except for two which quantify daytime frequency and nocturia separately with scores ranging from 0 to 4. A composite score between 10 and 14 indicates a strong diagnosis of IC/BPS with higher scores reflecting a greater degree of severity of symptoms and disease progressions as well as impact on quality of life.
Change in Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS) symptoms, as measured by the Global Response Assessment (GRA) | Baseline, Week 4, Week 8, Week 12, and Week 16
  The GRA is a single item, validated metric used to evaluate how ultimately effective a treatment method is from the perception of the patient. The GRA is structured on a 7-point scale centered at 0, indicating no change. The scales moves 3 points to the right of zero, indicating slight improvement, moderate improvement, and marked improvement, respectively, and 3 points to the left of zero, indicating slight worsening, moderate worsening, and marked worsening, respectively.
Change in Urinary symptoms, as measured by 3-day voiding diaries | Baseline, Week 4, Week 8, Week 12, and Week 16
  The voiding diary is a complete 3-day assessment of urinary symptoms (as they specifically pertain to IC/BPS) where patients themselves fill out quantitative and/or qualitative information in four categories at the time of each void: A) time of void, B) volume of voided urine (in mL) C) the severity of pain prior to void on a 0-10 numeric rating scale (NRS), D) the severity of pain 15 minutes after voiding on a 0-10 NRS, and E) time the participant went to bed at night and woke up in the morning. Following the completion of the 3-day voiding diary, the following four categories are calculated into quantifiable scores: 1) the total number of voids, 2) mean and total volume (in mL) of voided urine, 3) mean pre-voiding NRS pain score, and 4) mean post-voiding NRS score

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Walker, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van de Merwe JP, Nordling J, Bouchelouche P, Bouchelouche K, Cervigni M, Daha LK, Elneil S, Fall M, Hohlbrugger G, Irwin P, Mortensen S, van Ophoven A, Osborne JL, Peeker R, Richter B, Riedl C, Sairanen J, Tinzl M, Wyndaele JJ. Diagnostic criteria, classification, and nomenclature for painful bladder syndrome/interstitial cystitis: an ESSIC proposal. Eur Urol. 2008 Jan;53(1):60-7. doi: 10.1016/j.eururo.2007.09.019. Epub 2007 Sep 20. PMID 17900797
- [Background] Vasudevan V, Moldwin R. Addressing quality of life in the patient with interstitial cystitis/bladder pain syndrome. Asian J Urol. 2017 Jan;4(1):50-54. doi: 10.1016/j.ajur.2016.08.014. Epub 2016 Dec 2. PMID 29264207
- [Background] Keay SK, Birder LA, Chai TC. Evidence for bladder urothelial pathophysiology in functional bladder disorders. Biomed Res Int. 2014;2014:865463. doi: 10.1155/2014/865463. Epub 2014 May 8. PMID 24900993
- [Background] Parsons CL. The role of a leaky epithelium and potassium in the generation of bladder symptoms in interstitial cystitis/overactive bladder, urethral syndrome, prostatitis and gynaecological chronic pelvic pain. BJU Int. 2011 Feb;107(3):370-5. doi: 10.1111/j.1464-410X.2010.09843.x. Epub 2010 Dec 22. PMID 21176078
- [Background] Christmas TJ, Rode J, Chapple CR, Milroy EJ, Turner-Warwick RT. Nerve fibre proliferation in interstitial cystitis. Virchows Arch A Pathol Anat Histopathol. 1990;416(5):447-51. doi: 10.1007/BF01605152. PMID 2107633